CLINICAL TRIAL: NCT06099509
Title: Self-Administered 2-Hour Oral Glucose Tolerance Test: A Randomized Controlled Trial
Brief Title: Self-Administered 2-Hour Oral Glucose Tolerance Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2097104
Record Dates: First submitted 2023-10-18; First posted 2023-10-25 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Gestational Diabetes; Postpartum Disorder; Gestational Diabetes Mellitus in Pregnancy
MeSH Terms: conditions — Diabetes, Gestational; Puerperal Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-administered diabetes screen (Experimental): Self-administered 75-gram oral glucose tolerance test with 4-week virtual follow-up visit.
  Drug: GlucoCrush
  Interventions: Other: Self-administered oral glucose tolerance test
- Routine postpartum care (No Intervention): Office based oral glucose tolerance test at 6 weeks postpartum, per normal protocol.
  Drug: GlucoCrush

INTERVENTIONS:
Other: Self-administered oral glucose tolerance test — Participants will be asked to self-administer the postpartum 75-gram oral glucose tolerance test. They will be provided the glucose solution and instructions. A 4 week virtual visit will be arranged where the test results will be reported to the provider and appropriate follow up arranged based on the results of their screen.
  Arms: Self-administered diabetes screen

SUMMARY:
The goal of this randomized controlled trial is to evaluate whether self-administered postpartum diabetes screening tests in patients with gestational diabetes improves screening completion rates. The primary question it aims to answer is:

1. Does a self-administered 75-gram oral glucose tolerance test with virtual follow-up visit increase the rate of postpartum diabetes screening within 12 weeks of delivery?

DETAILED DESCRIPTION:
Gestational diabetes affects up to 10% of pregnancies, with increasing prevalence. Due to the risk of developing overt type 2 diabetes mellitus, patients are recommended to complete postpartum diabetes screening within 4-12 weeks of delivery. Despite these recommendations, screening rates remain low. Research evaluating reasons for low screening have identified social barriers like lack of transportation or childcare, as well as health literacy barriers. The consequences of missed screening include delay in diagnosis, delay in care, and ultimately higher health burden for the patient and the healthcare system.

This study seeks to evaluate a novel approach to increase uptake of recommended postpartum diabetes screening. The primary objective of this study is to determine if a self-administered postpartum diabetes screen (75-gram oral glucose tolerance test) increases screening completion rates. Our hypothesis is that the ability to perform the 75-gram oral glucose tolerance test at home will improve compliance with screening.

Additionally, we will evaluate the level of patient satisfaction with virtual follow-up in the intervention arm as a pre-specified additional outcome.

Eligible, consenting participants will be enrolled and randomized in a 1:1 ratio to the control arm (routine postpartum care with office-based diabetes screen) or intervention arm (self-administered diabetes screen). The randomization sequence will be generated by the study statistician using a block design. Investigators will remain masked to the randomization sequence.

All participants will be asked to complete a brief survey containing patient characteristics and two questions about perceived risk. Additional patient and neonatal data will be abstracted from the electronic medical record. All information will be stored in a secure password protected database.

Participants allocated to the intervention arm will receive the 75-gram oral glucose load and instructions prior to hospital discharge. The test should be administered approximately 4 weeks after delivery, and this date will be provided. They will be scheduled for a virtual visit approximately 4 weeks after delivery to report their results and discuss appropriate follow-up. Following this visit, participants will be asked to complete a modified version of the Telehealth Usability Questionnaire. The questionnaire contains five questions about their satisfaction with their telemedicine experience. The scoring is based on a likert scale, 1-7, with higher scores indicating higher satisfaction. If patients do not attend their 4-week virtual visit, they will be contacted one additional time to complete.

Participants will be scheduled for a routine 6-week postpartum visit.

Control arm participants will attend their routine 6-week postpartum visit where the postpartum diabetes glucose screen will be ordered. They can complete the test that day if they are fasting or will be responsible for arranging test completion on another day.

The study will conclude 12 weeks after delivery for each participant. At that time, any patients who have not completed the recommended postpartum diabetes screening will be contacted to ensure they have not completed screening outside of our health system/electronic medical record. If they are successfully contacted, they will be reported in intent-to-treat fashion based on self-reported completion of recommended screening.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age 18 years or older
* English or Spanish speaking
* Diagnosis of gestational diabetes with recommendation for postpartum screening, by any of the following criteria (1) HgbA1c 5.9-6.4% at ≤ 14 6/7 weeks, (2) HgbA1c ≥ 5.9% at 15-23 6/7 weeks, (3) 50-gram oral glucose tolerance test plasma glucose value ≥ 200 mg/dL, (4) 2 or more abnormal plasma glucose values on a 100-gram oral glucose tolerance test with the following thresholds: fasting ≥ 95 mg/dL, 1 hour ≥ 180 mg/dL, 2 hour ≥155 mg/dL, 3 hour ≥140 mg/dL or (5) fasting blood glucose ≥ 126
* No personal history of Type 1 or Type 2 diabetes defined by self-reported or documented history, or HgbA1c >/=6.5% at ≤ 14 6/7 weeks gestation
* Antepartum care with Prisma Health affiliated obstetric practices
* Delivery at Greenville Memorial Hospital
* Active Epic MyChart access at time of enrollment
* Capable of providing informed consent

Exclusion Criteria:

* Pre-pregnancy diagnosis of diabetes (Type 1, 2, or other form of diabetes)
* No glucometer or supplies for fingerstick glucose monitoring, or inability to perform fingerstick glucose monitoring
* Unable to provide informed consent
* Inability to follow up for routine postpartum care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Completion of 75-gram oral glucose tolerance test | within 12 weeks of delivery
  A comparison of the proportion of patients in each arm (intervention vs control) who complete recommended postpartum diabetes screening within 12 weeks of delivery. For the intervention arm, this will be completion of the self-administered 75-gram oral glucose tolerance test. For the control arm, this will be completion of the in-office 75-gram glucose tolerance test. The test will be considered completed in either arm if the patient has a fasting blood glucose >/=126 mg/dL (diagnostic of type 2 diabetes and does not require a post glucose load value), or both fasting and 2-hour post 75-gram glucose load blood glucose levels are documented.

OTHER OUTCOMES:
Patient satisfaction | within 12 weeks of delivery
  Patient satisfaction will only be assessed in the intervention arm. Satisfaction with their virtual visit will be assessed by evaluating scores from a modified version of the Telehealth Usability Questionnaire. This modified version contains 5 questions about satisfaction with telemedicine. The scoring is based on a likert scale, 1-7. 1 = strongly disagree, 7 = strongly agree, with higher scores indicating higher satisfaction.
  1. Telehealth improves my access to healthcare services.
  2. Telehealth provides for my healthcare need.
  3. Telehealth is an acceptable way to receive healthcare services.
  4. I would use telehealth services again.
  5. Overall, I am satisfied with this telehealth system.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Crockett, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Prisma Health/Greenville Memorial Hospital, Greenville, South Carolina, United States

REFERENCES:
- [Background] Quintanilla Rodriguez BS, Mahdy H. Gestational Diabetes. [Updated 2023 Aug 8]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2023 Jan-. Available from: https://www.ncbi.nlm.nih.gov/books/NBK545196/
- [Background] Blum AK. Insulin Use in Pregnancy: An Update. Diabetes Spectr. 2016 May;29(2):92-7. doi: 10.2337/diaspect.29.2.92. PMID 27182178
- [Background] "Gestational Diabetes Mellitus." ACOG Practice Bulletin, vol. 190, Feb. 2018, https://doi.org/https://www.acog.org/clinical/clinical-guidance/practice-bulletin/articles/2018/02/gestational-diabetes-mellitus.
- [Background] Tovar A, Chasan-Taber L, Eggleston E, Oken E. Postpartum screening for diabetes among women with a history of gestational diabetes mellitus. Prev Chronic Dis. 2011 Nov;8(6):A124. Epub 2011 Oct 17. PMID 22005617
- [Background] "Gestational Diabetes." Centers for Disease Control and Prevention, 2 Mar. 2022, www.cdc.gov/diabetes/basics/gestational.html#:~:text=Every%20year%2C%202%25%20to%2010,pregnancy%20and%20a%20healthy%20baby.
- [Background] Vounzoulaki E, Khunti K, Abner SC, Tan BK, Davies MJ, Gillies CL. Progression to type 2 diabetes in women with a known history of gestational diabetes: systematic review and meta-analysis. BMJ. 2020 May 13;369:m1361. doi: 10.1136/bmj.m1361. PMID 32404325
- [Background] Sinha DD, Williams RC, Hollar LN, Lucas HR, Johnson-Javois B, Miller HB, Stoermer A, Colditz GA, James AS, Herrick CJ. Barriers and facilitators to diabetes screening and prevention after a pregnancy complicated by gestational diabetes. PLoS One. 2022 Nov 18;17(11):e0277330. doi: 10.1371/journal.pone.0277330. eCollection 2022. PMID 36399472
- [Background] Dennison RA, Fox RA, Ward RJ, Griffin SJ, Usher-Smith JA. Women's views on screening for Type 2 diabetes after gestational diabetes: a systematic review, qualitative synthesis and recommendations for increasing uptake. Diabet Med. 2020 Jan;37(1):29-43. doi: 10.1111/dme.14081. Epub 2019 Jul 22. PMID 31317569
- [Background] Nielsen KK, Kapur A, Damm P, de Courten M, Bygbjerg IC. From screening to postpartum follow-up - the determinants and barriers for gestational diabetes mellitus (GDM) services, a systematic review. BMC Pregnancy Childbirth. 2014 Jan 22;14:41. doi: 10.1186/1471-2393-14-41. PMID 24450389